CLINICAL TRIAL: NCT02063724
Title: Pilot Phase I HER-2 Pulsed DC Vaccine to Prevent Recurrence for Patients With HER-2 Driven High Risk Invasive Breast Cancer
Brief Title: HER-2 Pulsed DC Vaccine to Prevent Recurrence of Invasive Breast Cancer
Acronym: Adjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-18777; 25113 (Other: CTSRMC, Abramson Cancer Center, University of Pennsylvania); NCT02110173 (obsolete NCT alias)
Record Dates: First submitted 2014-02-06; First posted 2014-02-14 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Invasive Breast Cancer; Breast Cancer; Immunotherapy; Vaccine; Dendritic Cell
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HER-2 Pulsed Dendritic Cell Vaccine (Experimental): 6 weekly HER-2 pulsed dendritic cell vaccines followed by 3 booster vaccines once every 3 months. Each dose will consist of between 1.0-2.0 x 10^7 cells and will be injected into 1-2 different normal groin lymph nodes or axillary nodes.
  Interventions: Biological: HER-2 pulsed Dendritic Cell Vaccine

INTERVENTIONS:
Biological: HER-2 pulsed Dendritic Cell Vaccine — 6 weekly HER-2 pulsed dendritic cell vaccines followed by 3 booster vaccines once every 3 months. Each dose will consist of between 1.0-2.0 x 10^7 cells and will be injected into 1-2 different normal groin lymph nodes or axillary nodes.

SUMMARY:
The purpose of this study is to determine the safety and immunogenicity of HER-2 pulsed DC1 vaccine in high risk HER-2 high and intermediate expression breast cancers. Participants will have HER-2 driven IBC at least Stage IIIA with N2 following chemotherapy with/without trastuzumab or recurrence exclusive of new primary tumor but rendered NED. Mammogram, laboratory studies, CT, and leukapheresis will be performed, in addition to vaccine administration.

DETAILED DESCRIPTION:
Dendritic cell cancer vaccines combined with chemotherapy may increase complete responses giving breast cancer specific immune cells greater opportunity to function while the immune repertoire is being shifted by chemotherapy to anti-breast cancer response and offer the chance to test secondary prevention of breast cancer in high risk settings. Participants with HER-2 driven IBC at least Stage IIIA with N2 (4 positive nodes) following chemotherapy with or without trastuzumab or those with recurrence exclusive of new primary tumor but rendered NED will be undergo mammograms, laboratory studies, and leukapheresis. Vaccines will be manufactured using participants' leukapheresis product, which will be administered in the Clinical Research Center 1 Dulles Building weekly for 6 weeks. Three booster vaccines will be administered at 3 month intervals following the initial induction vaccines. Immune analysis will be done after participant receives all induction vaccines and again after they receive all booster vaccines.

This study began at the Abramson Cancer Center of the University of Pennsylvania and will be continued at H. Lee Moffitt Cancer Center and Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Women over Age 18 years.
* Potential participants with Invasive Breast Cancer at least Stage IIIA, greater than or equal to N2 (>4 positive nodes) or have recurrent metastatic breast cancer rendered NED by any means that are classic HER-2 3+ 30%, 2+ IHC and FISH positive or HER-2 2+ FISH negative, that have completed chemotherapy and/or trastuzumab and are within 1 year from their last treatment and have no evidence of disease.
* Deemed to require anti-estrogen therapy for treatment of their breast cancer can continue anti-estrogen therapy during vaccinations.
* Women of childbearing age with a negative pregnancy test documented prior to enrollment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0 or 1.
* Willing to use birth control if necessary.
* Have voluntarily signed a written Informed Consent in accordance with institutional policies after its contents have been fully explained to them.

Exclusion Criteria:

* Pregnant or lactating.
* Positive for positive HIV or hepatitis C at baseline.
* Patients with coagulopathies, including thrombocytopenia with platelet count less than 75,000, INR greater than 1.5 and partial thromboplastin time greater than 50 sec.
* Major cardiac illness MUGA less than 50% EF.
* Pre-existing medical illnesses or medications which might interfere with the study as determined by Principal Investigator (PI).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2022-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Czerniecki, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Background] Czerniecki BJ, Roses RE, Koski GK. Development of vaccines for high-risk ductal carcinoma in situ of the breast. Cancer Res. 2007 Jul 15;67(14):6531-4. doi: 10.1158/0008-5472.CAN-07-0878. PMID 17638860
- [Background] Czerniecki BJ, Koski GK, Koldovsky U, Xu S, Cohen PA, Mick R, Nisenbaum H, Pasha T, Xu M, Fox KR, Weinstein S, Orel SG, Vonderheide R, Coukos G, DeMichele A, Araujo L, Spitz FR, Rosen M, Levine BL, June C, Zhang PJ. Targeting HER-2/neu in early breast cancer development using dendritic cells with staged interleukin-12 burst secretion. Cancer Res. 2007 Feb 15;67(4):1842-52. doi: 10.1158/0008-5472.CAN-06-4038. Epub 2007 Feb 9. PMID 17293384
- [Background] Koski GK, Koldovsky U, Xu S, Mick R, Sharma A, Fitzpatrick E, Weinstein S, Nisenbaum H, Levine BL, Fox K, Zhang P, Czerniecki BJ. A novel dendritic cell-based immunization approach for the induction of durable Th1-polarized anti-HER-2/neu responses in women with early breast cancer. J Immunother. 2012 Jan;35(1):54-65. doi: 10.1097/CJI.0b013e318235f512. PMID 22130160
- [Background] Sharma A, Koldovsky U, Xu S, Mick R, Roses R, Fitzpatrick E, Weinstein S, Nisenbaum H, Levine BL, Fox K, Zhang P, Koski G, Czerniecki BJ. HER-2 pulsed dendritic cell vaccine can eliminate HER-2 expression and impact ductal carcinoma in situ. Cancer. 2012 Sep 1;118(17):4354-62. doi: 10.1002/cncr.26734. Epub 2012 Jan 17. PMID 22252842
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled October 2014 through June 2017 at Abramson Cancer Center of the University of Pennsylvania and Moffitt Cancer Center.
Period: Overall Study
Arm/Group | HER-2 Pulsed Dendritic Cell Vaccine
Started | 15
Completed | 14
Not Completed | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Population: All participants.
Arm/Group | HER-2 Pulsed Dendritic Cell Vaccine
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 52 [30 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Rate of Treatment Regimen Completion
Description: Number of participants willing and able to complete treatment regimen, to address feasibility.
Time Frame: 12 months
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | HER-2 Pulsed Dendritic Cell Vaccine
Number analyzed (Participants) | 15
Participants | 14

2. Secondary Outcome: Immune Response
Description: Number of participants with immune response. Participants will undergo leukapheresis after completion of 6 vaccines and 3 boost vaccines for the purpose of obtaining lymphocytes and monocytes for in vitro immunologic testing.
Time Frame: 12 months
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | HER-2 Pulsed Dendritic Cell Vaccine
Number analyzed (Participants) | 15
Participants | 15

3. Secondary Outcome: Occurrence of Treatment Related Adverse Events
Description: Adverse Events reported as Related to Study Treatment, per adverse event category.
Time Frame: 2 years
Population: All participants.
Measure: Count of Participants; unit: Participants
Arm/Group | HER-2 Pulsed Dendritic Cell Vaccine
Number analyzed (Participants) | 15
Participants
  Rash | 1
  Citrate toxicity | 2
  Allergic reaction to pheresis | 1
  Tingling with pheresis | 1
  Fatigue | 1
  Chills | 2
  Fever | 2
  Bruising at site of injection | 1
  Lips and finger numbness and tingling | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | HER-2 Pulsed Dendritic Cell Vaccine
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 10/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HER-2 Pulsed Dendritic Cell Vaccine (N=15)
Hypertension (Vascular disorders) | 9 (15)
Axillary fullness (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Port infection (Infections and infestations) | 1 (1)
Cellulitis port site (Infections and infestations) | 1 (1)
Seizures (Nervous system disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Citrate toxicity (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (2)
Allergic reaction to pheresis (Immune system disorders) | 1 (1)
Tingling (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (3)
Chills (General disorders) | 2 (5)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (2)
Fever (General disorders) | 2 (2)
Bruising at site of injection (LEFT groin) (Injury, poisoning and procedural complications) | 1 (1)
Lip paresthesia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02063724/Prot_SAP_000.pdf